CLINICAL TRIAL: NCT03096483
Title: Clinical Evaluation of the OEC Elite Vascular Mobile Fluoroscopy System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor determination
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 104-2016-PTHS-0005
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Interventional Vascular Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- OEC Elite Imaging Arm (Experimental): Vascular, gastrointestinal (GI), urology or pain management procedures for which use of the OEC Elite system
  Interventions: Device: OEC Elite system

INTERVENTIONS:
Device: OEC Elite system — Adults undergoing vascular, gastrointestinal (GI), urology or pain management procedures

SUMMARY:
The purpose of the study is to collect survey data on the use of the OEC Elite Mobile Fluoroscopy System based on the routine clinical use of the device.

DETAILED DESCRIPTION:
This prospective clinical study is being conducted to acquire image guidance adequacy data from physicians conducting clinically-indicated vascular, gastrointestinal (GI), urology and pain management procedures for engineering use, as deemed appropriate by the Sponsor, for the investigational OEC Elite Mobile Fluoroscopy System (OEC Elite) in the vascular configuration. Clinical procedures included in this study will involve three (3) anatomical regions of interest - extremities and neck, thorax, and abdomen and pelvis. These regions are being targeted because they represent the range of clinical applications and anatomical regions intended for OEC Elite in the vascular configuration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 75 years (≥18 and ≤75 years old);
2. Clinical indication for a vascular, gastrointestinal (GI), urology or pain management procedure for which mobile fluoroscopy has been prescribed;
3. Able and willing to comply with study procedures; and
4. Able and willing to provide written informed consent to participate.

Exclusion Criteria:

1. Pregnant or suspected to be pregnant based on the opinion of and as documented by a medically qualified physician investigator;
2. Expected to be at increased risk due to study participation (e.g. due to allergies, sensitivities), in the medical opinion of an investigator; or
3. Previously participated in this study, or enrolled in another active GEHC study or other research study that could be expected to interfere with participation in study procedures, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Rapanos, Principal Investigator — Hamilton General Hospital
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OEC Elite Imaging Arm
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by site | 1

BASELINE CHARACTERISTICS:
Arm/Group | OEC Elite Imaging Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Imaging Guidance Adequacy Assessed by Number of Questionnaires
Description: Per-subject investigator report for procedure completion using the Investigational Device
Time Frame: 2 Months
Population: Excludes 1 (one) withdrawn subject because subject was withdrawn prior to study procedures using mobile fluoroscopy.
Measure: Number; unit: Image Guidance Adequacy Questionnaire
Arm/Group | OEC Elite Imaging Arm
Number analyzed (Participants) | 11
Image Guidance Adequacy Questionnaire | 11

2. Secondary Outcome: Number of Investigator Procedure Surveys Assessed by Survey Questionnaire
Description: The total number of per subject survey completion reflecting the investigator opinion of procedures completed with the investigational device
Time Frame: 2 months
Population: Excludes 1 (one) withdrawn subject because subject was withdrawn prior to study procedures using mobile fluoroscopy.
Measure: Number; unit: Procedure Survey Questionnaire
Arm/Group | OEC Elite Imaging Arm
Number analyzed (Participants) | 11
Procedure Survey Questionnaire | 11

ADVERSE EVENTS:
Time Frame: On a per-subject basis, from the point of enrollment to end of study procedure (i.e. approximately 0.5 days per subject).
Arm/Group | OEC Elite Imaging Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may not be used in future publications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03096483/Prot_SAP_000.pdf